CLINICAL TRIAL: NCT01193166
Title: A Twelve-Month, Prospective, Randomized, Active-Controlled, Open-Label, Flexible-Dose Study of Paliperidone Palmitate Compared With Oral Antipsychotic Treatment in Adults With Schizophrenia Who Have Been Recently Discharged From an Inpatient Psychiatric Hospital
Brief Title: Twelve Month Study Comparing Paliperidone Palmitate and Select Oral Antipsychotics in Adults With Schizophrenia Who Have Been Recently Discharged From an Inpatient Psychiatric Hospital
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: This study was stopped due to an internal reconsideration of priorities of the product portfolio.
Sponsor: Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CR017110; R092670SCH4003
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Risperdal; Paliperidone palmitate; Aripiprazole; Haloperidol; Olanzapine; Paliperidone; Perphenazine; Quetiapine
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate; Risperidone; Olanzapine; Aripiprazole; Quetiapine Fumarate; Perphenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- 001 (Experimental): paliperidone palmitate 78 117 156 or 234 mg monthly injection for 12 months
  Interventions: Drug: paliperidone palmitate
- 002 (Active Comparator): olanzapine flexible dosing as prescribed by the study doctor for 12 months
  Interventions: Drug: olanzapine
- 003 (Active Comparator): paliperidone flexible dosing as prescribed by the study doctor for 12 months
  Interventions: Drug: paliperidone
- 004 (Active Comparator): aripiprazole flexible dosing as prescribed by the study doctor for 12 months
  Interventions: Drug: aripiprazole
- 005 (Active Comparator): haloperidole flexible dosing as prescribed by the study doctor for 12 months
  Interventions: Drug: haloperidole
- 006 (Active Comparator): perphenazine flexible dosing as prescribed by the study doctor for 12 months
  Interventions: Drug: perphenazine
- 007 (Active Comparator): quetiapine flexible dosing as prescribed by the study doctor for 12 months
  Interventions: Drug: quetiapine
- 008 (Active Comparator): risperidone flexible dosing as prescribed by the study doctor for 12 months
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: paliperidone palmitate — 78, 117, 156, or 234 mg monthly injection for 12 months
  Arms: 001
Drug: risperidone — flexible dosing as prescribed by the study doctor for 12 months
  Arms: 008
Drug: olanzapine — flexible dosing as prescribed by the study doctor for 12 months
  Arms: 002
Drug: aripiprazole — flexible dosing as prescribed by the study doctor for 12 months
  Arms: 004
Drug: haloperidole — flexible dosing as prescribed by the study doctor for 12 months
  Arms: 005
Drug: quetiapine — flexible dosing as prescribed by the study doctor for 12 months
  Arms: 007
Drug: perphenazine — flexible dosing as prescribed by the study doctor for 12 months
  Arms: 006
Drug: paliperidone — flexible dosing as prescribed by the study doctor for 12 months
  Arms: 003

SUMMARY:
The study will assess the use of paliperidone palmitate compared with oral antipsychotic treatment in delaying time to a protocol-defined treatment failure over 12 months, in patients diagnosed with schizophrenia who were recently released from an inpatient psychiatric hospital.

DETAILED DESCRIPTION:
The primary objective of this study will be to compare paliperidone palmitate treatment with the randomly assigned oral antipsychotic treatment in delaying time to treatment failure over 12 months in subjects diagnosed with schizophrenia who were recently discharged from an inpatient psychiatric hospital. Patients will receive either paliperidone palmitate 78, 117, 156, or 234 mg monthly by injection for twelve months OR oral aripiprazole, haloperidol, olanzapine, paliperidone, perphenazine, quetiapine, and risperidone at doses selected by the study doctor.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to understand and sign the informed consent form approved by the Institutional Review Board (IRB)
* Must be an outpatient who, following an acute exacerbation of schizophrenia, has been discharged from an inpatient psychiatric hospital within 60 days of screening
* Have a current diagnosis of schizophrenia
* Have available a designated individual who is likely to have knowledge of the subject's health status and who agrees to let the study site personnel know of changes in the patient's circumstances
* Women must be postmenopausal (for at least 2 years), surgically sterile (hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy), abstinent, or if sexually active, be practicing a highly effective method of birth control

Exclusion Criteria:

* Allergies, hypersensitivity (anaphylaxis-type reaction), or intolerance to risperidone or paliperidone
* Actively abusing intravenous drugs
* Have a positive urine drug screen test for barbiturates, cocaine, amphetamines, or opiates at screening
* have an unstable medical illness
* Women who are pregnant or breast-feeding, or planning to become pregnant
* Have received injectable antipsychotic treatment within 2 injection cycles prior to screening
* Received treatment with clozapine within 3 months of screening
* Attempted suicide within 6 months before screening or are at imminent risk of suicide or violent behavior, as clinically assessed by the investigator at time of screening
* homeless at time of stuyd consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure defined as psychiatric hospitalization, suicide, discontinuation of treatment due to inadequate efficacy or safety/tolerability, treatment supplementation due to inadequate efficacy, or increase in psychiatric services | Up to 12 months

SECONDARY OUTCOMES:
Change in Clinical Global Impression-Severity score | Up to 12 months
Change in Global Assessment of Functionality score | Up to 12 months
Change in Medication Satisfaction Questionnaire score | Up to 12 months
Proportion of subjects with at least one psychiatric hospitalization | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Ortho-McNeil Janssen Scientific Affairs, LLC Clinical Trial, Study Director — Ortho-McNeil Janssen Scientific Affairs, LLC

REFERENCES:
- [Derived] Ibragimov K, Keane GP, Carreno Glaria C, Cheng J, Llosa AE. Haloperidol (oral) versus olanzapine (oral) for people with schizophrenia and schizophrenia-spectrum disorders. Cochrane Database Syst Rev. 2024 Jul 3;7(7):CD013425. doi: 10.1002/14651858.CD013425.pub2. PMID 38958149